CLINICAL TRIAL: NCT03114592
Title: Understanding the Role of Patient Behavior Change in Improving AKI Outcomes (Change AKI Study)
Brief Title: Understanding the Role of Patient Behavior Change in Improving AKI Outcomes
Acronym: Change AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00080287
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): * Complete a survey asking about kidney function and participant demographics.
  * Receive a one-month follow-up call (one month after hospital discharge date) and complete a phone survey about patient kidney function after discharge
- mHealth Tool (Experimental): * Complete a survey asking about kidney function and participant demographics.
  * Review a 15-20 minute educational tool on a tablet about kidney health
  * Receive a one-month follow-up call (one month after hospital discharge date) and complete a phone survey about patient kidney function after discharge
  Interventions: Other: mHealth tool

INTERVENTIONS:
Other: mHealth tool — The curriculum in the mHealth tool was derived in consultation with patient safety, informatics and adult educational curricula experts, and is comprised of clinical vignettes describing the post-hospital discharge stories of two hypothetical AKI survivors. opics of emphasis included NSAID risk awareness and avoidance of volume depletion when ill ("Sick Day Protocol").
  Arms: mHealth Tool

SUMMARY:
This study is looking to improve the safety of patients with acute kidney injury via education provided on a mobile tablet. This study will additionally examine if electronic tools, such as mobile tablets, can help.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an increasingly common complication of acute hospitalizations. Hospital-related AKI, commonly caused by hemodynamic changes or contrast exposure, carries a threat of adverse outcomes that persists following hospital discharge, with an independent and graded association with long-term mortality. It is estimated that, approximately 13% of individuals with acute coronary syndrome (ACS) will develop some degree of AKI during their hospitalization. Survivors of AKI consume significantly greater health resources than the general population, and suffer exceedingly poor renal outcomes, including persistent loss of kidney function, progression to end stage renal disease (ESRD), and increased risk of recurrent AKI. It is estimated that 25% of individuals with an AKI-related hospitalization will be readmitted with recurrent AKI within 12 months of discharge, highlighting a critical need to address ongoing AKI risk once the acute hospitalization is complete. Patient-centered educational interventions that intensify awareness of potentially hazardous situations may reduce AKI recurrence. For example, commonly prescribed therapies such as diuretics or ACE inhibitors may threaten the renal safety of individuals at high risk of recurrent AKI if taken when significantly volume deplete, such as during an acute gastroenteritis, and in most cases should be held until one can eat and drink normally; Nonsteroidal Anti-inflammatory Drugs (NSAIDs) may exacerbate AKI risk if taken in combination with diuretics or ACE inhibitors even when volume replete and should be completely avoided. Tailored educational curricula surrounding these and other topics pertinent to AKI survivors may reduce recurrent hospitalizations and lower healthcare costs. In the absence of a patient centered outpatient approach to AKI education, the development of effective and sustainable AKI prevention strategies remains unlikely.

Our long-term goal is to develop patient-centered educational materials to reduce AKI recurrence. We hypothesize that a tailored educational curriculum will improve patient awareness of potential hazards and reduce AKI recurrence among hospital-based AKI survivors. Therefore, our overall objective for this proposal is to pilot test and evaluate the feasibility of a patient-centered mobile health (mHealth) educational curriculum for hospitalized AKI survivors at Duke Medical Center.

Aim 1: To test the feasibility and acceptance of a mHealth patient safety curriculum in hospitalized AKI survivors.

Hypothesis 1: Patient safety risk awareness at 1 month will be higher in the educational intervention arm than the usual care arm.

Aim 2: To determine if a mHealth educational curriculum improves patient safety behaviors in AKI survivors.

Hypothesis 2: High-risk safety behaviors will be reduced at 1 month in AKI survivors receiving the educational intervention, but not in the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute kidney injury as diagnosed by renal care team
* On medical or surgical services
* Over 18 year of age
* Ability to read and speak English

Exclusion Criteria:

* Legal blindness or deafness
* Pregnant
* Cognitive impairment that limits ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Change in Patient Safety-Related Knowledge (Patient safety risk awareness) | Baseline, 1 month
  mHealth tool and how knowledge changes pre/post intervention
Change in Patient Safety Behavior and Risk awareness | Baseline, 1 month
  Survey assessing patient safety behavior and risk awareness

SECONDARY OUTCOMES:
User Satisfaction | 5 minutes
  Satisfaction of mHealth tool

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa J Diamantidis, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We are not sharing IPD